CLINICAL TRIAL: NCT07198399
Title: A Clinical Trial to Evaluate the Effects of a Supplement on Cognitive Health
Brief Title: Effects of Auri Super Mushroom Daily Gummies on Cognitive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auri Nutrition (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20739
Record Dates: First submitted 2025-09-14; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Decline; Focus Deficit
Keywords: Cognitive Health; Functional Mushrooms
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auri Cognitive Support Supplement (Experimental): Participants will take two Auri Super Mushroom Daily Gummies each morning for 8 weeks with their first meal and a glass of water.
  Interventions: Dietary Supplement: Auri Super Mushroom Daily Gummies

INTERVENTIONS:
Dietary Supplement: Auri Super Mushroom Daily Gummies — Each gummy contains a blend of 12 functional mushroom extracts (300 mg equivalent each).

SUMMARY:
This is a single-arm, open-label, virtual clinical trial evaluating the cognitive health effects of Auri Super Mushroom Daily Gummies in a population of 35 adult participants over 8 weeks. Participants will consume two gummies daily and complete validated cognitive testing and self-assessment questionnaires to assess changes in cognitive performance, energy, mood, memory, and overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female
* Be aged 30+
* Anyone who has been experiencing issues consistently for the last four weeks regarding all of the following:

Forgetfulness Inability to focus Low energy levels Low mood

* Anyone who is generally healthy - does not live with any uncontrolled chronic disease
* Willing to stop any other products or any medication or supplements that target cognition or cognitive health for the study duration
* Willing to maintain their current diet, sleep schedule, and activity level for the duration of the study
* Not undergone any surgeries or invasive treatments in the last six months
* Not had any major illness in the last three months
* Resides in the United States
* Not currently partaking in another research study and will not be partaking in any other research study for the next 8 weeks and at any point during this study's duration
* Willing to consult with their healthcare provider before enrolling in the study if taking any prescription medication

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Anyone with any allergies or sensitivities to any of the study product ingredients
* Anyone taking immunosuppressants
* Anyone taking blood thinners (anticoagulants)
* Any women who are pregnant, breastfeeding, or trying to conceive (or who will be at any point during the study period)
* Anyone unwilling to follow the study protocol
* Anyone with a history of substance abuse
* Anyone with intolerance or sensitivity to mushrooms

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Performance - Digit Span Test | Baseline, Week 2, Week 4, Week 6, and Week 8
  The Digit Span test measures working memory capacity. Participants are presented with a series of numbers and asked to recall them in order.
  Performance is scored based on the total number of correctly recalled sequences.
  Scale Name: Digit Span Score Range: 0 to 14 Direction: Higher scores indicate better cognitive performance.
Change in Cognitive Performance - Paired Associates Test | Baseline, Week 2, Week 4, Week 6, Week 8
  The Paired Associates task assesses memory by asking participants to recall which items were previously paired together.
  Score is based on the number of correct associations recalled.
  Scale Name: Paired Associates Score Range: 0 to 12 Direction: Higher scores indicate better cognitive performance.
Change in Attention and Processing Speed - Double Trouble Task | Baseline, Week 2, Week 4, Week 6, Week 8
  Double Trouble is a Stroop-like task that measures attention control and response inhibition.
  Performance is measured by accuracy (%) and completion time (seconds).
  Scale Name: Double Trouble Accuracy (%) Range: 0 to 100 Direction: Higher percentage indicates better attention and cognitive control.

SECONDARY OUTCOMES:
Self-Reported Focus - Questionnaire Score | Baseline, Week 2, Week 4, Week 6, and Week 8
  Participants rate their ability to focus using a Likert-style scale.
  Scale Name: Focus Rating Scale (1-10) Range: 1 (poor focus) to 10 (excellent focus) Direction: Higher scores indicate better focus
Self-Reported Memory - Questionnaire Score | Baseline, Week 2, Week 4, Week 6, and Week 8
  Participants self-assess memory retention using a 10-point Likert scale.
  Scale Name: Memory Rating Scale (1-10) Range: 1 (poor memory) to 10 (excellent memory) Direction: Higher scores indicate better memory

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States